CLINICAL TRIAL: NCT01412164
Title: A Prospective Multicenter Single-Arm Observational Registry Study Assessing the Safety and Efficacy of FIREHAWK Biodegradable Polymer Target-release Rapamycin-eluting Stent for the Treatment of Coronary Artery Disease: TARGET II
Brief Title: Observational Registry Study: FIREHAWK DES for Treating Coronary Artery Disease (CAD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TARGET II
Record Dates: First submitted 2011-08-05; First posted 2011-08-09 (Estimated); Results first posted 2016-03-17 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Coronary Artery Disease
Keywords: DES; CAD; FIREHAWK; MicroPort; PCI
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Firehawk (Experimental): Using Firehawk biodegradable polymer rapamycin-eluting stent for CAD
  Interventions: Device: FIREHAWK biodegradable polymer rapamycin-eluting stent

INTERVENTIONS:
Device: FIREHAWK biodegradable polymer rapamycin-eluting stent — DES PCI for CAD

SUMMARY:
The study aims to further assess the safety, efficacy and the performance of its delivery system of FIREHAWK rapamycin-eluting stent up to five years.

DETAILED DESCRIPTION:
This is a prospective open-labeled, multi-center, single-arm observational registry study. Approximately 1,100 subjects will be enrolled to evaluate the TLF as the primary endpoint at 12-month. Also, the study will follow up those subjects up to 5 years as the secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75, male or unpregnant women
* Evidence of non-symptomatic ischemia, stable or non-stable angina or past MI
* Native coronary artery target lesion
* Target lesion length <=60mm, target lesion vessel diameter 2.25mm-4.0mm
* Target lesion diameter stenosis>=70%
* For each target lesion, Firehawk stent implantation only
* Understand the study purpose, willing to participate and sign the letter of consent
* Acceptance of clinical follow-up

Exclusion Criteria:

* Acute MI within 72 hours
* Unprotected LM and intervention-required three-vessel lesions
* Calcified lesion failed in pre-dilation and twisted lesion
* Bridge vessel lesion
* Any stent implanted within one year
* Severe heart failure (HYHA>=III) or LVEF<40%
* Renal deficiency, blood creatinine > 2.0mg/dl
* Bleeding tendency
* Allergic to aspirin, clopidogrel, ticlopidine, dye, rapamycin and metal
* Life expectation <12 months
* History of not achieving study finish
* No compliances to the protocol
* Heart implantation subjects

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2011-08; Primary Completion 2013-02 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Runlin Gao, M.D., Prof., Principal Investigator — Fu Wai Hospital, Beijing, China
Locations (1):
- Fuwai Hospital, Beijing, China

REFERENCES:
- [Derived] Gao Z, Zhang R, Xu B, Yang Y, Ma C, Li H, Chen S, Han Y, Yuan Z, Lansky AJ, Guan C, Leon MB, Gao R; TARGET Investigators. Safety and efficacy of a novel abluminal groove-filled biodegradable polymer sirolimus-eluting stent for the treatment of de novo coronary lesions: two-year results from a prospective patient-level pooled analysis of TARGET trials. Catheter Cardiovasc Interv. 2015 Mar;85 Suppl 1:734-43. doi: 10.1002/ccd.25861. Epub 2015 Feb 19. PMID 25678281

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Firehawk
Started | 730
Completed | 683
Not Completed | 47

BASELINE CHARACTERISTICS:
Arm/Group | Firehawk
Number analyzed (Participants) | 730
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.71 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 213
  Male | 517
Region of Enrollment [Number; unit: participants]
  China | 730

OUTCOME MEASURES:

1. Primary Outcome: TLF (Target Lesion Failure) Rate
Description: Percentage of participants with determination of TLF ,TLF is the composite of cardiac death, target vessel MI and clinically driven TLR
Time Frame: 12 months after index procedure
Measure: Number; unit: percentage of participants with TLF
Arm/Group | Firehawk
Number analyzed (Participants) | 730
percentage of participants with TLF | 4.4

2. Secondary Outcome: Stent Implantation Success Rate (SIS Rate)
Description: Stent implantation success (SIS) means participant successfully implanted stent, defined as residual stenosis of the lesion less than 30% and TIMI bloodflow Grade III
Time Frame: immediately after the procedure
Measure: Number; unit: percentage of participants with SIS
Arm/Group | Firehawk
Number analyzed (Participants) | 730
percentage of participants with SIS | 96.8

3. Secondary Outcome: Patient-related Cardiovascular Clinical Composite Endpoints
Description: Participants with cardiovascular clinical composite endpoints. Cardiovascular clinical composite endpoints defined as the composite of all death, all MI and vascular reconstruction.
Time Frame: 1 years after index PCI
Measure: Count of Participants; unit: Participants
Arm/Group | Firehawk
Number analyzed (Participants) | 730
Participants | 46

4. Secondary Outcome: Patient-related Cardiovascular Clinical Composite Endpoints
Description: as for outcome 3
Time Frame: 3 years after index PCI
Measure: Count of Participants; unit: Participants
Arm/Group | Firehawk
Number analyzed (Participants) | 712
Participants | 77

5. Secondary Outcome: Patient-related Cardiovascular Clinical Composite Endpoints
Description: as for outcome 3
Time Frame: 5 years after index PCI
Measure: Count of Participants; unit: Participants
Arm/Group | Firehawk
Number analyzed (Participants) | 683
Participants | 112

6. Secondary Outcome: TLF (Target Lesion Failure)
Description: as for outcome 1
Time Frame: 1 years after index PCI
Measure: Number; unit: percentage of participants with TLF
Arm/Group | Firehawk
Number analyzed (Participants) | 730
percentage of participants with TLF | 4.38

7. Secondary Outcome: TLF (Target Lesion Failure)
Description: Participants with the determination of TLF, TLF is the composite of cardiac death, target vessel MI and clinically driven TLR
Time Frame: 3 years after index PCI
Measure: Count of Participants; unit: Participants
Arm/Group | Firehawk
Number analyzed (Participants) | 712
Participants | 46

8. Secondary Outcome: TLF (Target Lesion Failure)
Description: Participants with the determination of TLF. TLF is the composite of cardiac death, target vessel MI and clinically driven TLR at 12 months post procedure
Time Frame: 5 years after index PCI
Measure: Count of Participants; unit: Participants
Arm/Group | Firehawk
Number analyzed (Participants) | 683
Participants | 59

ADVERSE EVENTS:
Arm/Group | Firehawk
All-Cause Mortality (participants affected / at risk) | 30/683
Serious Adverse Events (participants affected / at risk) | 112/683
Other Adverse Events (participants affected / at risk) | 0/730
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Firehawk (N=683)
Perioperative myocardial infarction (Cardiac disorders) | 38
Target lesion revascularization (Cardiac disorders) | 67
Death (Psychiatric disorders) | 30
Definite/probable in-stent thrombosis (Cardiac disorders) | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Firehawk (N=730)
Arrhythmia (Cardiac disorders) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No